CLINICAL TRIAL: NCT00989196
Title: Clinical Study to Investigate the Pharmacokinetics, Efficacy, Safety and Immunogenicity of Human-cl rhFVIII, a Newly Developed Human Cell-line Derived Recombinant FVIII Concentrate in Previously Treated Patients With Severe Hemophilia A
Brief Title: Clinical Study to Investigate the Pharmacokinetics, Efficacy, Safety and Immunogenicity of a Recombinant FVIII in Patients With Severe Hemophilia A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GENA-01
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Results first posted 2014-01-17 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human-cl rhFVIII (Experimental)
  Interventions: Biological: Human-cl rhFVIII
- Kogenate FS (Active Comparator)
  Interventions: Biological: Kogenate FS

INTERVENTIONS:
Biological: Human-cl rhFVIII — 50 IU/kg for PK dose
  Arms: Human-cl rhFVIII
Biological: Kogenate FS — 50 IU/kg for PK dose
  Arms: Kogenate FS

SUMMARY:
This is a clinical study to investigate the pharmacokinetics, efficacy, safety and immunogenicity of human-cl rhFVIII, a newly developed human cell-line derived recombinant FVIII concentrate in previously treated patients with severe Hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A (FVIII:C <= 1%)
* Male subjects between 12 and 65 years of age
* Body weight 25 kg to 110 kg
* Previously treated with FVIII concentrate for at least 150 EDs

Exclusion Criteria:

* Other coagulation disorder than hemophilia A
* Present or past FVIII inhibitor activity

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sigurd Knaub, PhD, Study Director — Octapharma
Locations (9):
- United States (6):
  - UCLA Orthodpedic Hospital, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of Colorado, Denver, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - RUSH University Medical Center, Chicago, Illinois
  - University of Medicine and Dentistry, New Brunswick, New Jersey
- Prof. Lissitchkov, Sofia, Bulgaria
- Germany (2):
  - Medizinische Hochschule, Hanover, Lower Saxony
  - Vivantes Klinikum, Berlin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in the USA, 2 centers in Germany and 1 center in Bulgaria. The first patient was included on May 27, 2010 and the last patient finished the study on September 18, 2012
Pre-assignment Details: The patients started the study with a PK period. The PK period had a cross-over design (Kogenate vs Human cl rhFVIII) and subjects received either Kogenate first and Human cl rhFVIII second or vice versa. Once the PK measure had been done, the patient started the treatment period with Human cl rhFVIII only.
Groups:
- Human c1 rhFVIII First Crossover, Then Treatment: Participants were randomized to receive Human-cl rhFVIII (50 IU/kg bodyweight) first, then Kogenate FS (50 IU/kg bodyweight)second in the Crossover period. In the Treatment Period, participants received Kogenate (50 IU/kg bodyweight)
- Kogenate First Crossover, Then Treatment: Participants were randomized to receive Kogenate (50 IU/kg) first (14 days), then Human-cl rhFVIII (50 IU/kg bodyweight) second (14 days) in the Crossover period. In the Treatment Period, participants received Human-cl rhFVIII (50 IU/kg bodyweight)
Period: PK Crossover Period
Arm/Group | Human c1 rhFVIII First Crossover, Then Treatment | Kogenate First Crossover, Then Treatment
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0
Period: Treatment Period
Arm/Group | Human c1 rhFVIII First Crossover, Then Treatment | Kogenate First Crossover, Then Treatment
Started | 10 | 12
Completed | 9 | 12
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Human cl rhFVIII: Human-cl rhFVIII and Kogenate in cross-over design:50 IU/kg for PK dose
Arm/Group | Human cl rhFVIII
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 10
  Bulgaria | 6
  Germany | 6

OUTCOME MEASURES:

1. Primary Outcome: The Area Under the Concentration Curve for Human-cl rhFVIII Compared to Kogenate FS
Description: After the infusion of 50IU/kg bw of Human-cl rhFVIII and Kogenate FS respectively, FVIII activity levels were measured at various time points before and after the infusion. FVIII level results derived from the chromogenic FVIII assay were used to calculate the mean of the area under the curve normalized to the dose administered.
Time Frame: At baseline (prior to infusion), 0.25, 0.5, 0.75, 1, 3, 6, 9, 12, 24, 30 and 48 hours after the end of the infusion.
Measure: Mean (Standard Deviation); unit: h IU/mL (IU/kg)
Groups:
- Human cl rhFVIII: Human-cl rhFVIII 50 IU/kg for PK dose
- Kogenate FS: Kogenate FS 50 IU/kg for PK dose
Arm/Group | Human cl rhFVIII | Kogenate FS
Number analyzed (Participants) | 22 | 22
h IU/mL (IU/kg) | 0.39 (0.14) | 0.38 (0.09)
Statistical Analysis 1: Comparison: Human cl rhFVIII vs Kogenate FS; Test type: Non-Inferiority or Equivalence — For the comparison of the PK profile of Human-cl rhFVIII with Kogenate, the 90% confidence intervals for the ratio or log-ratio of Human-cl rhFVIII over Kogenate for selected, dose independent or dose adjusted, PK parameters will be presented. In addition a formal statistical procedure will test whether the ratio of mean AUCs is within a 80 to 125% range to show bioequivalence; Ratio = 0.98, 90% CI 2-sided [0.874 to 1.107]

2. Secondary Outcome: Invivo Half-life (T1/2) for Human-cl rhFVIII Compared to Kogenate FS
Description: as for outcome 1
Time Frame: At baseline (prior to infusion), 0.25, 0.5, 0.75, 1, 3, 6, 9, 12, 24, 30 and 48 hours after the end of the infusion.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Human cl rhFVIII | Kogenate FS
Number analyzed (Participants) | 22 | 22
hours | 14.73 (9.96) | 16.14 (5.88)

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Human-cl rhFVIII Compared to Kogenate FS
Description: as for outcome 1
Time Frame: At baseline (prior to infusion), 0.25, 0.5, 0.75, 1, 3, 6, 9, 12, 24, 30 and 48 hours after the end of the infusion.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Human cl rhFVIII | Kogenate FS
Number analyzed (Participants) | 22 | 22
IU/mL | 1.462 (0.223) | 1.394 (0.2)

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) for Human-cl rhFVIII Compared to Kogenate FS
Description: as for outcome 1
Time Frame: At baseline (prior to infusion), 0.25, 0.5, 0.75, 1, 3, 6, 9, 12, 24, 30 and 48 hours after the end of the infusion.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Human cl rhFVIII | Kogenate FS
Number analyzed (Participants) | 22 | 22
hours | 0.35 (0.23) | 0.34 (0.2)

5. Secondary Outcome: Mean Residence Time (MRT) for Human-cl rhFVIII Compared to Kogenate FS
Description: as for outcome 1
Time Frame: At baseline (prior to infusion), 0.25, 0.5, 0.75, 1, 3, 6, 9, 12, 24, 30 and 48 hours after the end of the infusion.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Human cl rhFVIII | Kogenate FS
Number analyzed (Participants) | 22 | 22
hours | 19.45 (12.02) | 20 (5.61)

6. Secondary Outcome: Volume of Distribution at Steady State (Vss) for Human-cl rhFVIII Compared to Kogenate FS
Description: as for outcome 1
Time Frame: At baseline (prior to infusion), 0.25, 0.5, 0.75, 1, 3, 6, 9, 12, 24, 30 and 48 hours after the end of the infusion.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Human cl rhFVIII | Kogenate FS
Number analyzed (Participants) | 22 | 22
mL/kg | 49.58 (17.27) | 53.32 (13.57)

7. Secondary Outcome: Clearance (CL) for Human-cl rhFVIII Compared to Kogenate FS
Description: as for outcome 1
Time Frame: At baseline (prior to infusion), 0.25, 0.5, 0.75, 1, 3, 6, 9, 12, 24, 30 and 48 hours after the end of the infusion.
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Human cl rhFVIII | Kogenate FS
Number analyzed (Participants) | 22 | 22
mL/h/kg | 2.94 (1.18) | 2.75 (0.64)

8. Secondary Outcome: Efficacy of On-demand Treatment of Bleeding Episodes
Description: After each infusion of IMP and at the end of a BE, the following efficacy assessment is made by the subject (together with the Investigator in case of on-site treatment):
  Excellent: Abrupt pain relief and/or unequivocal improvement in objective signs of bleeding within approximately 8 hours after a single infusion.
  Good: Definite pain relief and/or improvement in signs of bleeding within approximately 8 - 12 hours after an infusion requiring up to 2 infusions for complete resolution.
  Moderate: Probable or slight beneficial effect within approximately 12 hours after the first infusion requiring more than two infusions for complete resolution.
  None: No improvement within 12 hours, or worsening of symptoms, requiring more than 2 infusions for complete resolution.
  The assessment was made at the end of a BE in case more than one infusion was needed.
Time Frame: From 1st treatment after PK cycle 2 until study end.
Measure: Number; unit: percentage of bleeding episodes
Units Other Than Participants: Bleeding episodes
Arm/Group | Human cl rhFVIII
Number analyzed (Participants) | 22
Number analyzed (Bleeding episodes) | 986
percentage of bleeding episodes
  Excellent | 60.3
  Good | 34.1
  Moderate | 5.5
  None | 0

9. Secondary Outcome: Immunogenicity (Number of Patients That Developed an Inhibitor During the Course of the Study)
Description: Inhibitor activity was determined by the modified Bethesda assay (Nijmegen modification) at study entry, then immediately before both PK cycles, in the 48 hour sample of both PK cycles, after 10 to 15 EDs with human-cl rhFVIII, at the 3-month visit (± 2 weeks), then every 3 months (± 2 weeks) until study completion, and after >50 EDs (except for some patients who may finish the study before they achieve 50 EDs), with human-cl rhFVIII (i.e. at the study completion visit).
Time Frame: study entry, then immediately before both PK cycles, in the 48 hour sample of both PK cycles, after 10 to 15 EDs with human-cl rhFVIII, at the 3-month visit (± 2 weeks), then every 3 months (± 2 weeks) until study completion, and after >50 EDs (except for
Measure: Number; unit: participants
Arm/Group | Human cl rhFVIII
Number analyzed (Participants) | 22
participants | 0

ADVERSE EVENTS:
Time Frame: From 27 May 2010 to 18 September 2012 (study end)
Description: All Adverse events were collected regardless of the intervention. Kogenate is a licensed product and the active ingredient is the same as for the investigational product Human cl rhFVIII. Therefore no distinction was made whether an AE occurred after Kogenate or after Human cl rhFVIII administration.
Groups:
- Human cl rhFVIII and Kogenate FS: All participants. Human-cl rhFVIII and Kogenate in cross-over design:50 IU/kg for PK period. After the PK period all participants received Human-cl rhFVIII in the treatment period.
Arm/Group | Human cl rhFVIII and Kogenate FS
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 6/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human cl rhFVIII and Kogenate FS (N=22)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1)
DEPRESSION SUICIDAL (Psychiatric disorders) | 1 (1)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human cl rhFVIII and Kogenate FS (N=22)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Protein urine present (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Octapharma agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Octapharma supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial. Octapharma also reserves the right to review data prior to publishing and provide comments/changes within a certain time period.